CLINICAL TRIAL: NCT06853353
Title: Nurse-led Consultations in Heart Failure Within the 'FIL-EAS' Evaluation and Support Care Pathway for Heart Failure Patients
Acronym: ISPIC FILEAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CHITS-017
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; Nurse; Heart Failure Nurse Specialists; Advanced practice nursing; Treatment titration; Care pathway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic heart failure receiving consultations from a Heart Failure Specialist Nurse.
  Interventions: Other: Heart Failure Specialist Nurses consultations

INTERVENTIONS:
Other: Heart Failure Specialist Nurses consultations — Heart Failure Specialist Nurses consultations

SUMMARY:
The management of chronic heart failure, following current guidelines, requires the implementation and adjustment of therapies to limit mortality and morbidity associated with disease progression. However, this period of treatment titration remains challenging due to the need for multiple, closely spaced consultations. The difficulty in maintaining this consultation frequency, coupled with the current decline in medical demographics, largely explains the lack of treatment titration or even initiation and the existing therapeutic inertia. Concurrently, medical telemonitoring is emerging as an essential tool in heart failure management, offering significant benefits for both patients and healthcare professionals.

In this context, new forms of nursing practices have emerged, such as advanced practice nursing, aimed at improving the care of patients with chronic diseases. However, only limited data are currently available regarding the functioning and impact of these consultations in France.

The "Evaluation and Support Pathway for Heart Failure Patients (FIL-EAS ic)" has systematically integrated this new model of consultations provided by heart failure nurse specialists. Given their significant and growing role within the pathway, it appears necessary to thoroughly evaluate these consultations to propose improvements and maximize their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or over
* Patient seen in nurse-led consultations for heart failure between January 1, 2023 and December 31, 2023

Exclusion Criteria:

* Patient opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient seen in nurse-led consultations for heart failure between January 1, 2023 and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Type of consultation | 1-year period
  Medical telemonitoring, treatment titration, advanced practice nurse follow-up
Patient's medical history | 1-year period
  Patient's clinical characteristics will be analyzed : number and type of medical histories
Treatments implemented | 1-year period
  Type and dose of treatment initiated for heart failure will be analyzed.
Number of consultations | 1-year period
  The number of consultations will be analyzed by type of activity (medical telemonitoring, treatment titration, advanced practice nurse follow-up).
Number of hospitalizations | 1-year period
  The number of hospitalizations and re-hospitalizations during the 12 months of follow-up will be analyzed.

SECONDARY OUTCOMES:
Type of referral | 1-year period
  The type of referral will be analyzed : in-hospital (cardiology or non-cardiology) or out-of-hospital (cardiologist, general practitioner, private nurse or Advanced Practice Registered Nurse)
Reason for discontinuation of titration consultation | 1-year period
  The reason for the discontinuation of titration consultations will be analyzed.
Left ventricular ejection fraction (LVEF) | 1-year period
  Echocardiography data during therapy titration will be analyzed.
Modification of recommended treatment doses | 1-year period
  Modification of recommended treatment doses in heart failure will be analyzed in the overall cohort and according to the level of LVEF at initial management.
Rate of detection of iron deficiency | 1-year period
  The rate of detection of iron deficiency will be analyzed according to whether or not Ferinject supplementation is used.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde LE CAIGNEC, Nurse, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer; Jocelyne CANDEL, Advanced Practice Nurse, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France